CLINICAL TRIAL: NCT03356080
Title: Clinical Efficacy and Safety of DLAAG Protocol in the Treatment of Refractory/Relapse of Acute Myeloid Leukemia (AML) and Myelodysplastic Syndrome With Blast Excess: a Multicenter, Single-arm, Prospective Clinical Study
Brief Title: DLAAG in the Treatment of Acute Myeloid Leukemia (AML) and Myelodysplastic Syndrome With Blast Excess
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Tong Ren Hospital (Other)
Responsible Party: Principal Investigator, Liu Ligen, head of hematology department, Shanghai Tong Ren Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DLAAG
Record Dates: First submitted 2017-11-09; First posted 2017-11-29 (Actual); Last update posted 2017-11-29 (Actual); Status verified 2017-11

CONDITIONS: Acute Myeloid Leukemia; Myelodysplastic Syndrome
Keywords: decitabine; retinoid acid; cytarabine C; Granulocyte Colony Stimulating Factor; acute myeloid leukemia; Myelodysplastic Syndrome
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes | interventions — Decitabine; Cytarabine; Granulocyte Colony-Stimulating Factor; Filgrastim

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DLAAG (Experimental): All patients receive 1-2 cycles of induction chemotherapy,that is DLAAG,which is expected to be 6 weeks/cycle,including decitabine,cytarabine, all-transretinoic acid,and Granulocyte Colony-Stimulating Factor(G-CSF).
  patients with CR after the first course of induction therapy (DLAAG) will continue to receive 1 cycle of consolidation therapy, while those with therapy failure will continue the second course of induction therapy. If CR is not achieved, quit the study.
  Patients who achieve CR after induction therapy will be in accordance with the guidelines, such as the proposed active treatment of allogeneic hematopoietic stem cell transplantation
  Interventions: Drug: Decitabine; Drug: Cytarabine; Drug: All-transretinoic acid; Drug: G-CSF

INTERVENTIONS:
Drug: Decitabine — Decitabine,iv,0.1-0.2mg/kg, Day1-Day3 per week,up to 3 weeks
  Other Names: Qingweike
Drug: Cytarabine — cytarabine, iv,15mg/m2 q12h, Day1-Day10
  Other Names: Cytosar
Drug: All-transretinoic acid — All-transretinoic acid, 45mg/d Day4-Day6;15mg/d Day7-Day20
  Other Names: Ailike
Drug: G-CSF — G-CSF 300ug,sc,Day 0 until CR is achieved
  Other Names: Filgrastim

SUMMARY:
The purpose of this study is to evaluate of the clinical efficacy and safety of DLAAG protocol in the treatment of acute myeloid leukemia (AML) and myelodysplastic syndrome with blast excess

ELIGIBILITY:
Inclusion Criteria:

1. corresponding to the AML (except M3) or high-risk MDS diagnostic criteria, with any of the following circumstances:

   ①secondary AML patients (including AML secondary to MDS)

   ②corresponding to refractory AML diagnostic standard ( relapsed refractory acute myeloid leukemia Chinese guidelines(2017 Edition): Refractory AML diagnostic criteria: invalid after standard treatment 2 cycles of untreated cases; consolidation therapy after CR and then recurrence within 12 months; recurrence after 12 months and then invalid after conventional chemotherapy ; relapse of ≥ 2 times ; extramedullary leukemia continued existence.

   ③corresponding to recurrent AML diagnostic criteria (relapsed refractory acute myeloid leukemia China guidelines (2017 Edition): peripheral blood leukemia cells or bone marrow progenitor cells appear again > 0.050 after CR (with the exception of bone marrow regeneration after consolidation chemotherapy and other reasons) or leukemia cells infiltration appear in extramedullary

   ④corresponding to MDS refractory anemia with blasts excess (RAEB) diagnosis standards
2. Age ≥18 years old
3. Eastern Cooperative Oncology Group(ECOG) score 0-3
4. Expected survival ≥8 weeks
5. Patients must be able to understand and be willing to participate in this study, and signed informed consent

Exclusion Criteria:

1. acute promyelocytic leukemia (M3 type)
2. Other types of MDS patients except RAEB
3. with other advanced malignant tumors
4. patients with uncontrolled severe infection, and can not tolerate chemotherapy with other serious underlying diseases
5. patients with heart failure: ejection fraction (EF) < 30%, New York Heart Association(NYHA) standard, cardiac insufficiency in class II or above

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2017-07-07 (Actual); Primary Completion 2019-07-07 (Estimated); Study Completion 2020-07-07 (Estimated)

PRIMARY OUTCOMES:
Complete Response Rate (CR) | at the end of every course(about 4 weeks)
  Morphologic CR - patient independent of transfusions
  * Absolute neutrophil count(ANC) >1000/ Microliter(mcL)
  * Platelets ≥100,000/mcL
  * No residual evidence of extramedullary disease
  Cytogenetic CR - cytogenetics normal (in those with previously abnormal cytogenetics)
  Molecular CR - molecular studies negative
  CR with incomplete blood cells count recovery(CRi) - There are some clinical trials, particularly those that focus on the elderly or those with antecedent myelodysplasia, that include a variant of complete response referred to as CRi. This has been defined as <5% marrow blasts, either ANC <1000/mcL or platelets <100,000/mcL, and transfusion independence but with persistence of cytopenia (usually thrombocytopenia).

SECONDARY OUTCOMES:
Early death rate | the death rate after treating Day1 to Day30
  The rate of early death within 30 days
Leukemia free survival (LFS) | from enrolling to the end of 2-year following up
  Morphologic leukemia-free state Bone marrow <5% blasts in an aspirate with spicules No blasts with Auer rods or persistence of extramedullary disease
Overall survival(OS) | from enrolling to the end of 2-year following up
  The time from the date of enrolling to the date of death due to any reasons or the last following date
The rate of adverse reaction the rate of adverse reaction | from enrolling to the end of 2-year following up
  the rate of adverse reaction, according to Standard for World Health Organization(WHO) acute and subacute toxicity
Duration of hospitalization | from enrolling to the end of 2-year following up
  The time from the date of be hospitalized to the date of be discharged
The rate of relapse | from enrolling to the end of 2-year following up
  Relapse following complete response is defined as reappearance of leukemic blasts in the peripheral blood or the finding of more than 5% blasts in the bone marrow, not attributable to another cause (eg, bone marrow regeneration after consolidation therapy) or extramedullary relapse

CONTACTS AND LOCATIONS:
Overall Officials: Ligen Liu, Principal Investigator — Shanghai Tong Ren Hospital
Locations (6):
- China (6):
  - Beijing Friendship Hospital, Beijing
  - Fujian Medical University Union Hospital, Fuzhou
  - The People's Hospital of Guangxi Zhuang Autonomous Region, Nanning
  - Shanghai Tong Ren hospital, Shanghai
  - The center hospital of Shanghai Fengxian District, Shanghai
  - First Affiliated Hospital of Zhengzhou University., Zhengzhou